CLINICAL TRIAL: NCT00776373
Title: A Phase I/II, Open-label Single Institution Study Evaluating Rapamycin in Combination With High-dose Etoposide and Cytarabine in Relapsed or Refractory Aggressive Lymphoid Malignancies
Brief Title: Rapamycin in With High-Dose Etoposide and Cytarabine in Relapsed/Refractory Aggressive Lymphoid Malignancies
Acronym: UPCC 25406
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 25406
Record Dates: First submitted 2008-10-19; First posted 2008-10-21 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: ALL; Burkitt's Lymphoma; Lymphoblastic Leukemia; CML
Keywords: ALL; Burkitt's Lymphoma; Adult T-Cell leukemia/lymphoma; Lymphoblastic leukemia; CML in lymphoid blast crisis patients; HiVAC; Rapamycin
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Sirolimus; Etoposide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental): Rapamycin in combination with High Dose Etoposide and Cytarabine (HiVAC)
  Interventions: Drug: Rapamycin; Drug: High dose etoposide and cytarabine (HiVAC)

INTERVENTIONS:
Drug: Rapamycin — Rapamycin,by mouth, loading dose followed by a single daily dose for 8 days (dose level 1 = load of 9 mg followed by 3 mg daily doses, dose level 2 = 12 mg with daily doses of 4 mg
Drug: High dose etoposide and cytarabine (HiVAC) — Etoposide 500 mg/m2/day IV and Cytarabine 2000 mg/m2/day IV every 24 hours for 4 days.

SUMMARY:
Assess the safety, tolerability and efficacy of rapamycin in combination with HiVAC in relapsed and refractory patients with aggressive lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Advanced lymphoid leukemia (primary refractory ALL; Relapsed ALL; CML in lymphoid accelerated phase or blast crisis; relapsed or refractory Burkitt's lymphoma; relapsed or refractory T-cell adult leukemia/lymphoma; relapsed or refractory lymphoblastic lymphoma
* >= 18 and <= 65 years of age ECOG performance status 0, 1 Life expectancy >= 4 weeks Able to consume oral medication Required initial laboratory values: Creatinine <= 2.0mg/dL, total or direct bilirubin <= 1.5 mg/dL, SGPT(ALT) <=ULN, glucose < 200 mg/dL, negative pregnancy test for women with child bearing potential

Exclusion Criteria:

* Subjects must not be receiving any chemotherapy agents (except Hydroxyurea)
* Subjects must not have received high-dose Ara-C within 6 months of relapse
* Subjects must not be receiving growth factors, except for erythropoietin
* No currently active second malignancy other than non-melanoma skin cancers
* No subjects with uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, MI within the last 6 months or serious uncontrolled cardiac arrhythmia
* Subjects taking Carbamazepine, Rifabutin, Rifampin, Rifapentine, St. John's wort, Clarithromycin, Cyclosporine, Diltiazem, Erythromycin, Telithromycin, Verapamil, Tacrolimus
* Known HIV positivity or AIDS-related illness
* Evidence of cerebellar dysfunction or prior history of cerebellar dysfunction with Ara-C administration
* Pregnant or lactating
* Uncontrolled infection
* Taking fluconazole, voriconazole, itraconazole and ketoconazole currently or within one week of study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-01; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability and efficacy of rapamycin in combination with HiVAC in relapsed and refractory patients with aggressive lymphoid malignancies | Study completion

SECONDARY OUTCOMES:
Assess and quantify phosphorylation of p70S6 kinase | Study completion
Whether increased mTOR pathway inhibition correlates with response to therapy with rapamycin and HiVAC | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Selina Luger, MD, Principal Investigator — University of Pennsylvania Abramson Cancer Center
Locations (1):
- University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania, United States